CLINICAL TRIAL: NCT07024264
Title: Caloric Estimation Using Predictive Equations and Indirect Calorimetry in ICU Patients
Brief Title: Measured Versus Estimated Energy Requirement in the ICU Patients
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202409050
Record Dates: First submitted 2025-05-14; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-10

CONDITIONS: Critical Illness; Energy Requirement; Equation; Indirect Calorimetry; Malnutrition
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Total energy requirement calculated by predictive equation — Critically ill patients are highly susceptible to malnutrition, making accurate caloric estimation essential to prevent both underfeeding and overfeeding during the acute phase in the ICU. Although predictive equations (PE) are widely used to estimate energy requirement, indirect calorimetry (IC) remains the gold standard. This study aimed to compare energy requirements estimated by PE and IC across different BMI categories.

SUMMARY:
The goal of this observational study is to compare energy requirements estimated by predictive equation and indirect calorimetry across different BMI categories, and to examine how these estimates, along with early nutritional strategies and progressive caloric delivery relate to ICU outcomes. The main questions it aims to answer are:

1. To evaluate whether predictive equation and/or indirect calorimetry provides accurate caloric targets in critically ill patients.
2. To identify high-risk malnutrition patients (underweight, normal and overweight, obese) who may benefit most from IC-based measurement.
3. To investigate the impact of caloric strategies and nutritional achievement during the acute phase on the length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Length of ICU stay > 4 days
* Mechanically ventilated adults (>20 y/o)
* Tube feeding
* At high risk of malnutrition by Global Leadership Initiative on Malnutrition (GLIM) criteria: underweight and obesity
* Doctor's preference: cachexia, hypermetabolic status, TPN etc.,…

Exclusion Criteria:

* Length of ICU stay <4 days
* Mechanically ventilated adults (<=20 y/o)

Ages: 20 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU and ventilator dependent in Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome was ICU length of stay. | From admitted to ICU which defined as day 1, until transferred to the general wards or expired, up to 12 weeks.
  This study aimed to compare energy requirements estimated by PE and IC across different BMI categories, and to examine how these estimates, along with early nutritional strategies and progressive caloric delivery relate to the length of ICU stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Background] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Background] De Waele E, Jonckheer J, Wischmeyer PE. Indirect calorimetry in critical illness: a new standard of care? Curr Opin Crit Care. 2021 Aug 1;27(4):334-343. doi: 10.1097/MCC.0000000000000844. PMID 33990505
- [Background] Zusman O, Theilla M, Cohen J, Kagan I, Bendavid I, Singer P. Resting energy expenditure, calorie and protein consumption in critically ill patients: a retrospective cohort study. Crit Care. 2016 Nov 10;20(1):367. doi: 10.1186/s13054-016-1538-4. PMID 27832823